CLINICAL TRIAL: NCT06836401
Title: Effect of Topical Metronidazole in Reducing Periodontal Probing Depth: A Split Mouth Clinical Trial
Brief Title: Topical Metronidazole vs Control in Reducing Periodontal Pockets in a Split Mouth Clinical Trial
Acronym: Perio_topic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, JAVIER MONTERO, Head of the Department of Surgery, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USAL_Nº201700008745
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Periodontal Disease; Periodontal Inflammation
Keywords: periodontal pocket; periodontal disease; periodontal inflammation
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket | interventions — Dental Scaling; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metronidazole (Experimental): These periodontal pockets will be treated with a metronidazole-based gel
  Interventions: Procedure: Root scaling; Drug: Topical Gel
- Carbopole (Sham Comparator): These deep periodontal pockets (>4mm) are treated with a placebo gel made of carbopol gel
  Interventions: Procedure: Root scaling; Drug: Topical Gel

INTERVENTIONS:
Procedure: Root scaling — Scaling and root planing is a deep cleaning below the gumline used to remove plaque and tartar that cover the root in the periodontal pockets. This intervention is carried out in both control and experimental sites
Drug: Topical Gel — A gel (experimental: metronidazole VS control: carbopol) is introduced in the recently cleaned periodontal pocket. The allocation of either experimental or control gel was distributed randomly, being masked both the patient and the clinician.

SUMMARY:
The effect of both the mechanical treatment and the topical metronidazol in reduccing the inflammation and depth of the periodontal pockets were assessed on the first bicuspids.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal patients with all first premolars suffering from moderate periodontal pockets (>4mm of probing depth)

Exclusion Criteria:

* No patients received antibiotics nor periodontal treatment in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Probing depth | Both one month and three months after root scaling
  Probing depth is assessed at 6 points around the first bicuspids (mesiovestibular, midvestibular, distovestibular, mesiolingual, midlingual, distolingual)
Mieloperoxidase ng/mL | Both one and three months after root scaling
  The determination of the quantity of mieloperoxidase ng/mL was assessed from the crevicular fluid of the treated bicuspids

CONTACTS AND LOCATIONS:
Overall Officials: Javier Montero, Main Researcher, Principal Investigator — University of Salamanca
Locations (1):
- Dental School of the Faculty of Medicine, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided
This work is planned to be a PhD dissertation and we are not sure if sharing data would hamper the originality of the future thesis